CLINICAL TRIAL: NCT06153030
Title: Unexpected Diagnosis in Right Lower Quadrant Pain: Right Colon Diverticulitis
Status: Completed | Type: Observational
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Naz Tayyar, Resident Medical Doctor, Haydarpasa Numune Training and Research Hospital
Other Study IDs: Haydarpasa Numune Training and
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Diverticulitis, Colonic
Keywords: acute diverticulitis; right colon; emergency; pain
MeSH Terms: conditions — Diverticulitis, Colonic; Emergencies; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with right colonic diverticulitis
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
BACKGROUND: Acute right lower quadrant pain is a common symptom in emergency departments. The most common etiology is thought to be acute appendicitis. Other etiologies may be overlooked. Acute right colon diverticulitis is one of them. It is usually seen in male and young patients. It is more common in Asian population and rare in Western countries. Ultrasonography (USG) and computed tomography (CT) are used for radiologic diagnosis.

OBJECTIVES: The aim of this study was to investigate the diagnosis, treatment and surgical management of right colon diverticulitis.

DETAILED DESCRIPTION:
DESIGN: Retrospective cross-sectional analysis SETTING: Research and training hospital (Tertiary care center) In our study, patients hospitalized in our hospital clinic between 2018 and 2022 with the diagnosis of right colon diverticulitis were retrospectively analyzed. Age, gender, WSES grade, whether surgery was performed or not, laboratory values, iv antibiotherapies given, length of hospitalization and mortality were evaluated.

MAIN OUTCOME MEASURES: The CRP, the need for surgical intervention vs conservative treatment .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with right colonic diverticulitis

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with right colonic diverticulitis between the years of 2018-2022
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
The need for surgical intervention | time frame is the length of stay usually between 1-14 days
  The patients were followed up conservatively if they had their diagnosis in the acute settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner GA, O'Grady MJ, Purcell RV, Frizelle FA. The Epidemiology and Etiology of Right-Sided Colonic Diverticulosis: A Review. Ann Coloproctol. 2021 Aug;37(4):196-203. doi: 10.3393/ac.2021.00192.0027. Epub 2021 Jul 21. PMID 34284562
- [Background] Papatriantafyllou A, Dedopoulou P, Soukouli K, Karioris I, Tsochatzis S. Right-Sided Diverticulitis: A Rare Cause of Right-Sided Abdominal Pain. Cureus. 2023 Apr 4;15(4):e37123. doi: 10.7759/cureus.37123. eCollection 2023 Apr. PMID 37153306
- [Background] Ma Z, Liu W, Zhou J, Yao L, Xie W, Su M, Yang J, Shao J, Chen J. Management and long-term outcomes of acute right colonic diverticulitis and risk factors of recurrence. BMC Surg. 2022 Apr 7;22(1):132. doi: 10.1186/s12893-022-01578-z. PMID 35392887
- [Background] Kahveci S, Tokmak TT, Yildirim A, Mavili E. Acute right-sided colonic diverticulitis mimicking appendicitis: a report of two cases. J Clin Ultrasound. 2013 May;41(4):238-41. doi: 10.1002/jcu.21967. Epub 2012 Aug 1. PMID 22855407
- [Background] Shin JH, Son BH, Kim H. Clinically distinguishing between appendicitis and right-sided colonic diverticulitis at initial presentation. Yonsei Med J. 2007 Jun 30;48(3):511-6. doi: 10.3349/ymj.2007.48.3.511. PMID 17594161
- [Background] Lee JH, Ahn BK, Lee KH. Conservative treatment of uncomplicated right-sided diverticulitis: a systematic review and meta-analysis. Int J Colorectal Dis. 2021 Aug;36(8):1791-1799. doi: 10.1007/s00384-021-03913-x. Epub 2021 Mar 25. PMID 33765173
- [Background] Park SM, Kwon TS, Kim DJ, Lee YS, Cheung DY, Oh ST, Kim JG, Lee IK. Prediction and management of recurrent right colon diverticulitis. Int J Colorectal Dis. 2014 Nov;29(11):1355-60. doi: 10.1007/s00384-014-1938-3. Epub 2014 Jul 6. PMID 24997717
- [Background] Park HC, Kim BS, Lee K, Kim MJ, Lee BH. Risk factors for recurrence of right colonic uncomplicated diverticulitis after first attack. Int J Colorectal Dis. 2014 Oct;29(10):1217-22. doi: 10.1007/s00384-014-1941-8. Epub 2014 Jul 1. PMID 24980689
- [Background] Kim YC, Chung JW, Baek JH, Lee WS, Kim D, Park YH, Yang JY, Lee WK. Risk Factors for Recurrence of Right Colonic Diverticulitis. Dig Surg. 2019;36(6):509-513. doi: 10.1159/000494297. Epub 2018 Nov 8. PMID 30408791
- [Background] Kim MR, Kye BH, Kim HJ, Cho HM, Oh ST, Kim JG. Treatment of right colonic diverticulitis: the role of nonoperative treatment. J Korean Soc Coloproctol. 2010 Dec;26(6):402-6. doi: 10.3393/jksc.2010.26.6.402. Epub 2010 Dec 31. PMID 21221240
- [Background] Lee KY, Lee J, Park YY, Oh ST. Routine colonoscopy may be needed for uncomplicated acute right colonic diverticulitis. BMC Gastroenterol. 2021 Feb 27;21(1):91. doi: 10.1186/s12876-021-01672-1. PMID 33639847
- [Result] Huang SS, Sung CW, Wang HP, Lien WC. The outcomes of right-sided and left-sided colonic diverticulitis following non-operative management: a systematic review and meta-analysis. World J Emerg Surg. 2022 Nov 1;17(1):56. doi: 10.1186/s13017-022-00463-7. PMID 36320045
- [Result] Palacios Huatuco RM, Pantoja Pachajoa DA, Liano JE, Picon Molina HA, Palencia R, Doniquian AM, Parodi M. Right-sided acute diverticulitis in the West: experience at a university hospital in Argentina. Ann Coloproctol. 2023 Apr;39(2):123-130. doi: 10.3393/ac.2021.00402.0057. Epub 2021 Nov 24. PMID 34814235
- [Result] Oh MY, Shin R, Heo SC, Lim HK, Kim MJ, Park JW, Ryoo SB, Jeong SY, Park KJ. Investigation of the clinical features and recurrence patterns of acute right-sided colonic diverticulitis: A retrospective cohort study. Ann Med Surg (Lond). 2022 Aug 18;81:104431. doi: 10.1016/j.amsu.2022.104431. eCollection 2022 Sep. PMID 36147058
- [Result] Rov A, Ben-Ari A, Barlev E, Pelcman D, Susmalian S, Paran H. Right-sided diverticulitis in a Western population. Int J Colorectal Dis. 2022 Jun;37(6):1251-1256. doi: 10.1007/s00384-022-04135-5. Epub 2022 May 4. PMID 35505198